CLINICAL TRIAL: NCT06541522
Title: Impact of Belt Position on the Results of PEEP Titration by Electrical Impedance Tomography During Acute Respiratory Distress Syndrome
Brief Title: Impact of Belt Position on the Results of PEEP Titration by EIT During ARDS
Acronym: REPEIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REPEIT
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: ARDS
Keywords: ARDS; mechanical ventilation; EIT

STUDY DESIGN:
Intervention Model Description: Once the patient is included in the research, two PEEP titrations monitored by EIT will be performed, each with the electrode belt positioned at a different chest height. The order will be drawn at random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEP titrations (Other)
  Interventions: Device: EIT

INTERVENTIONS:
Device: EIT — Two PEEP titrations monitored by EIT will be performed, each with the electrode belt positioned at a different chest height (2nd intercostal space or 5th intercostal space). The order will be drawn at random.

SUMMARY:
ARDS is a frequent reason for hospitalization in intensive care. In order to improve its management, doctors seek to limit the mechanical ventilation-induced injuries (VILI) that can occur. PEEP is a parameter that plays a role in the appearance of VILI, and its adjustment can be optimized by EIT. The EIT is a non-invasive, non-irradiating, real-time monitoring device, today widely used for the optimization of ventilation in patients intubated for ARDS. The positioning of the EIT belt at different chest heights could influence the result of the PEEP titration.

DETAILED DESCRIPTION:
The aim of this study is to test the hypothesis that the position (2nd intercostal space or 5th intercostal space) of the EIT (Electrical Impedance Tomography) belt significantly influences the result of PEEP (Positive Expiratory Pressure) titration.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of moderate to severe ARDS (PaO2/FiO2 ratio ≤ 200 mmHg) within 72 hours following intubation
* Criteria for moderate to severe ARDS for less than 72 hours
* Passive ventilation in controlled assisted ventilation (no spontaneous ventilation)
* Consent of next of kin

Exclusion Criteria:

* Age < 18 years
* ECMO
* Pneumothorax
* Pacemaker or implantable defibrillator
* Chest trauma in the last 3 months
* Skin peeling (Burned, Lyell)
* Intracranial hypertension
* Uncontrolled shock (noradrenaline >5 mg/h)
* Pregnant woman
* Adult patient protected within the meaning of the law
* Lack of social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Impact of the position of the electrode belt on the results of PEEP titration by EIT. | Day 0
  Optimal PEEP determined by PEEP titration using the crossing point method.

SECONDARY OUTCOMES:
Impact of the existence of intra-tidal recruitment on the discordance between PEPEIT and PEPCRS | Day 0
  Variability of the impedance variation during insufflation of the tidal volume ("tidal impedance variation) during titration measured by the relative interquartile coefficient (Q3-Q1)/median
Factors associated with a discordance between PEPEIT and PEPCRS | Day 0
  Variability of the impedance variation during insufflation of the tidal volume ("tidal impedance variation) during titration measured by the relative interquartile coefficient (Q3-Q1)/median
Discrepancy between compliance measured according to impedance and compliance measured according to exhaled volume | Day 0
  Regional ventilation delay (RVD)